CLINICAL TRIAL: NCT01461837
Title: Familial Haploidentical T-Cell Depleted Transplantation in High-Risk Sickle Cell Disease (IND 14359)
Brief Title: Haplo T-Cell Depleted Transplantation in High-Risk Sickle Cell Disease
Acronym: HaploSCD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: UCSF Benioff Children's Hospital Oakland (Other); Medical College of Wisconsin (Other); Washington University School of Medicine (Other); Tufts Medical Center (Other); University of California, San Francisco (Other); University of California, Los Angeles (Other); Miltenyi Biomedicine GmbH (Industry); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC526-4090; FD-R-0004090 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2011-10-19; First posted 2011-10-28 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; stem cell transplantation; haploidentical
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Haplo Stem Cell Transplantation (Experimental): CD34 selected T-cell depleted allogeneic SCT
  Interventions: Drug: CD34 selected T-cell depleted allogeneic SCT

INTERVENTIONS:
Drug: CD34 selected T-cell depleted allogeneic SCT — Hydroxyurea (60 mg/kg/day) and azathioprine (3 mg/kg/day) day -59 to day -11; fludarabine (30 mg/m2) Days -17, -16, -15, -14, -13; busulfan (3.2 mg/kg/day) Days -12, -11, -10, -9; thiotepa (10 mg/kg IV) day -8; cyclophosphamide (50 mg/kg) Days -7, -6, -5, -4; TLI on day -3; rabbit ATG (2.0 mg/kg/day) day -5,-4,-3, and -2; Stem Cell infusion day 0
  Other Names: Familial haploidentical; T-cell depleted; allogeneic stem cell transplantation; high risk Sickle Cell Disease

SUMMARY:
This study is being done to determine the safety and outcome (long-term control) of a high-dose chemotherapy regimen followed by an infusion of CD34 selected (immune cells) stem cells from a partially matched adult family member donor, called haploidentical stem cell transplantation, in high-risk sickle cell disease patients.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
The purpose of this study is to investigate host myeloimmunosuppressive conditioning followed by familial haploidentical T cell depleted allogeneic stem cell transplantation in patients with high risk Sickle Cell Disease (SCD). It is hypothesized that it will be safe and well tolerated, and result in sustained donor chimerism, acceptable engraftment and immune reconstitution. Also, that it will limit SCD related organ damage resulting in improved and/or stable neurological, neurocognitive, pulmonary and pulmonary vascular function and health related quality of life (QOL).

Patients 2-20.99 years of age with a diagnosis of high-risk SCD and with an unaffected HLA partially matched family donor and meeting eligibility criteria (inclusion and exclusion criteria) are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous Hemoglobin S Disease, or Hemoglobin S Beta0/+ thalassemia
* Patients must demonstrate one or more of the following Sickle Cell Disease Complications

  1. Clinically significant neurologic event (stroke) or any neurologic deficit lasting >24 hours that is accompanied by an infarct on cerebral MRI
  2. Minimum of two episodes of acute chest syndrome.
  3. Recurrent painful events (at least 3 in the 2 years prior to enrollment).
  4. Abnormal TCD study requiring starting on chronic transfusion therapy.
  5. At least one silent infarct lesion on a MRI scan of the head.
* A familial haploidentical donor without homozygous sickle cell disease
* Adequate organ function (renal, liver, cardiac and pulmonary function)
* Karnofsky or Lansky (age appropriate) Performance Score ≥50%
* Liver biopsy is optional to assess for iron overload in chronically transfused patients.

Exclusion Criteria:

* Females who are pregnant or breast-feeding
* SCD Patients with documented uncontrolled infection
* SCD patients who have an unaffected HLA matched family donor willing to proceed to donation
* Karnofsky/Lansky (age appropriate) Performance Score <50% (hemiplegia alone secondary to a previous stroke is not an exclusion)
* Demonstrated lack of compliance with medical care.
* Clinically significant fibrosis or cirrhosis of the liver
* Previously received a HSCT

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2012-01; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Treatment related events | 1 year
  Death, primary or late graft rejection, or recurrence of disease and acceptable rate of hematopoietic engraftment, acute and chronic graft-versus-host disease

SECONDARY OUTCOMES:
neurological/neurocognitive status | 2 years
  Change from baseline in neurological/neurocognitive status
Pulmonary/pulmonary vascular status | 2 years
  Change from baseline of Pulmonary/pulmonary vascular status
Health-related quality of life | 4 years
  Change from baseline of Health-related quality of life (CHRIs-HSCT/CHRIs-General)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — New York Medical College
Locations (6):
- United States (6):
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Lurie Children's Hospital, Chicago, Illinois
  - Washington University/St. Louis Children's Hospital, St Louis, Missouri
  - New York Medical College, Valhalla, New York
  - Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Braniecki S, Vichinsky E, Walters MC, Shenoy S, Shi Q, Moore TB, Talano JA, Parsons SK, Flower A, Panarella A, Fabricatore S, Morris E, Mahanti H, Milner J, McKinstry RC, Duncan CN, van de Ven C, Cairo MS. Neurocognitive outcome in children with sickle cell disease after myeloimmunoablative conditioning and haploidentical hematopoietic stem cell transplantation: a non-randomized clinical trial. Front Neurol. 2024 May 22;15:1263373. doi: 10.3389/fneur.2024.1263373. eCollection 2024. PMID 38841694
- [Derived] Parsons SK, Rodday AM, Weidner RA, Morris E, Braniecki S, Shenoy S, Talano JA, Moore TB, Panarella A, Flower A, Milner J, Fabricatore S, Mahanti H, van de Ven C, Shi Q, Cairo MS. Significant improvement of child physical and emotional functioning after familial haploidentical stem cell transplant. Bone Marrow Transplant. 2022 Apr;57(4):586-592. doi: 10.1038/s41409-022-01584-y. Epub 2022 Feb 2. PMID 35110690
- See also: Consortium website for Parent-to-Child (haplo) Bone Marrow Transplant for Sickle Cell Disease (SCD) — http://www.sicklecelltransplantconsortium.org/